CLINICAL TRIAL: NCT07335471
Title: A Comprehensive Intervention Program for Preventing Cardiovascular and Cerebrovascular Complications in Uremic Patients on Maintenance Hemodialysis
Brief Title: Prevention and Management of Cardiovascular and Cerebrovascular Complications in Maintenance Hemodialysis (MHD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Municipal Hospital of Anhui Province (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SZH-CVRP-2023-01
Record Dates: First submitted 2025-12-16; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Uremia; Chronic; Cardiovascular Diseases (CVD); Cerebrovascular Disorders; Intradialytic Hypotension; Ultrafiltration Intolerance; Dialysis Adequacy
MeSH Terms: conditions — Uremia; Bronchiolitis Obliterans Syndrome; Cardiovascular Diseases; Cerebrovascular Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Continuous High-Glucose Infusion (Other)
  Interventions: Other: Continuous High-Glucose Infusion and Regular Hemoperfusion in Maintenance Hemodialysis

INTERVENTIONS:
Other: Continuous High-Glucose Infusion and Regular Hemoperfusion in Maintenance Hemodialysis — hemoperfusion

SUMMARY:
Background and Purpose: This clinical study aims to explore and validate two innovative treatment strategies to address two major challenges faced by patients on maintenance hemodialysis (uremia): the high incidence of cardiovascular and cerebrovascular complications and the common occurrence of ultrafiltration intolerance/refractory intradialytic hypotension.

Study Design: The research consists of two main parts, employing a prospective, interventional design.

Hemoperfusion (HP) for Cardiovascular/Cerebrovascular Complications: The investigators plan to enroll approximately 200 uremic patients on dialysis at the study center. Initially, a detailed survey of their existing cardiovascular health status and related risk factors will be conducted. Subsequently, a standardized hemoperfusion treatment platform will be established and evaluated, observing its effects on removing relevant toxins and improving biochemical markers. Finally, a subset of patients who have already developed such complications will be invited to participate in a comparative study. They will be randomly assigned to receive either conventional dialysis or conventional dialysis combined with intensified hemoperfusion therapy to systematically assess the efficacy and safety of the combined regimen.

Continuous High-Glucose Infusion for Ultrafiltration Intolerance: For patients suffering from severe ultrafiltration intolerance and refractory hypotension during glucose-free dialysis that does not respond to standard therapies (36 patients have been enrolled), an interventional study was conducted. Patients received a continuous infusion of 50% glucose solution during dialysis, supplemented by glucose boluses as needed. The study primarily observed whether this protocol could safely extend dialysis duration, increase ultrafiltration volume, and improve dialysis adequacy and related symptoms.

Participants: The study will be conducted at the Blood Purification Center of Suzhou Hospital. The main participants are adults aged 18 or older, diagnosed with uremia and receiving maintenance hemodialysis. For the cardiovascular/cerebrovascular part, patients must meet specific inclusion criteria; for the ultrafiltration intolerance part, patients must be diagnosed with refractory intradialytic hypotension unresponsive to standard therapy.

Study Procedures: All participants will provide informed consent before joining the study. The study will collect patient medical history, conduct physical examinations, blood tests, and questionnaires according to the protocol. Patients receiving hemoperfusion or high-glucose infusion interventions will undergo close monitoring of vital signs and efficacy evaluations before and after treatment. Some participants may be scheduled for regular follow-up to understand their long-term outcomes.

Potential Benefits and Risks: Participants may benefit directly from the study, for example: through the new treatment strategies, they may achieve better control of cardiovascular risks, reduce discomfort associated with hypotension (such as dizziness and cramping), and increase ultrafiltration volume and adequacy per session, potentially improving quality of life and long-term health outcomes. The risks involved are primarily routine medical risks associated with hemoperfusion or intravenous glucose infusion, such as bleeding or infection at the puncture site, blood glucose fluctuations, etc. All procedures will be performed by experienced medical staff under strict supervision to maximize patient safety.

Social Significance: The results of this study are expected to provide clinicians with new, evidence-based treatment options for managing the complex and challenging complications in uremic dialysis patients. If proven effective and safe, these protocols may be incorporated into clinical practice guidelines, helping more patients achieve adequate and comfortable dialysis, ultimately improving patient prognosis and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80 years.
2. Receiving maintenance hemodialysis (MHD) for 3 months or longer.
3. Diagnosis of severe ultrafiltration intolerance (UFI), defined as either:

   Persistent pre-dialysis hypotension (systolic blood pressure <100 mmHg), OR

   Recurrent intradialytic hypotension (IDH), defined per KDOQI guidelines as a decrease in systolic blood pressure to <90 mmHg or by >20 mmHg from baseline, accompanied by symptoms.
4. Failure to achieve target ultrafiltration volume (mean UFV <1.5 L per session) despite at least 4 weeks of conventional interventions (e.g., dialysate cooling, sodium profiling, sequential ultrafiltration).
5. Inadequate dialysis delivery, defined as a mean single-pool Kt/V of less than 1.2.

Exclusion Criteria:

1. Acute infection, myocardial infarction, or major surgery within the past 3 months.
2. Uncontrolled diabetes mellitus, defined as a glycated hemoglobin (HbA1c) level greater than 9%.
3. Severe liver dysfunction (Child-Pugh class C).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-07-20 (Actual)

PRIMARY OUTCOMES:
Incidence of Intradialytic Hypotension (IDH) Events | 2 years
  This primary outcome measure assesses the frequency of intradialytic hypotension events during hemodialysis sessions. IDH is strictly defined as a systolic blood pressure drop of ≥20 mmHg or a mean arterial pressure drop of ≥10 mmHg, accompanied by clinical symptoms (e.g., dizziness, nausea, cramps) requiring nursing intervention. The measure will be reported as the number of IDH events per patient per dialysis session, calculated from nursing records and continuous blood pressure monitoring data throughout the intervention period.
Dialysis Adequacy Measured by Single-Pool Kt/V | 2 years
  This measure assesses the efficacy of solute clearance during hemodialysis using the single-pool Kt/V formula, which is calculated based on pre- and post-dialysis blood urea nitrogen levels, dialysis duration, and ultrafiltration volume. A higher Kt/V value indicates more adequate dialysis.
Dialysis Adequacy Measured by Urea Reduction Ratio (URR) | 2 years
  This measure assesses dialysis efficacy by the percentage reduction of blood urea nitrogen during a treatment session. URR is calculated from pre- and post-dialysis urea nitrogen levels. It is reported as a percentage (%).
Serum B-type Natriuretic Peptide (BNP) Level | 2 years
  This measure evaluates the change in cardiac load and fluid status by assessing serum BNP concentration. Blood samples will be collected at baseline and post-intervention for analysis. It is reported in picograms per milliliter (pg/mL).
Serum Levels of Phosphate, Calcium, and Intact Parathyroid Hormone (iPTH) | 2 years
  This measure evaluates changes in mineral and bone metabolism. Fasting blood samples will be collected at baseline and at scheduled intervals during the intervention period. Serum phosphate and calcium levels will be measured using standard laboratory biochemical analyzers, reported in mmol/L. Serum iPTH level will be measured using electrochemiluminescence immunoassay, reported in pg/mL.
Severity of Uremic Pruritus | 2 years
  This measure assesses the intensity of dialysis-related itch. The severity of pruritus will be evaluated by patients using a validated Visual Analogue Scale (VAS), ranging from 0 (no itch) to 10 (worst imaginable itch). The assessment will be recorded weekly during dialysis sessions throughout the study period. The outcome will be reported as the mean VAS score.
Treatment Failure Rate for Refractory Ultrafiltration Intolerance | 2 years
  This measure evaluates the clinical efficacy in managing ultrafiltration intolerance. Treatment failure is operationally defined as the inability to complete the prescribed dialysis duration or to achieve the target ultrafiltration volume due to intradialytic hypotension (IDH) that is unresponsive to the study's glucose infusion protocol, necessitating early session termination. This binary outcome (Yes/No) will be determined per dialysis session based on nursing and medical records.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Emergent Adverse Events as Assessed by CTCAE v5.0 | 2 years
  All adverse events occurring from the start of the study intervention until the end of follow-up will be recorded. Each event will be graded for severity and assessed for relationship to the study procedures according to the Common Terminology Criteria for Adverse Events version 5.0.
Incidence of Acute Platelet Count Reduction and Periprocedural Hypersensitivity Reactions during Hemoperfusion | 2 years
  Two specific procedure-related events will be monitored: 1) Acute platelet reduction: defined as a decrease in platelet count by >30% from the pre-hemoperfusion value measured within 24 hours post-procedure. 2) Hypersensitivity reaction: defined as the occurrence of symptoms such as rash, hypotension, bronchospasm, or anaphylaxis during or within 2 hours after the hemoperfusion procedure.
Peak Intradialytic Blood Glucose Level and Change in Pre-dialysis Fasting Glucose | 2 years
  Glucose levels will be monitored to assess metabolic perturbation. 1) Peak intradialytic glucose: the highest capillary blood glucose value (in mmol/L) recorded during any dialysis session with glucose infusion. 2) Fasting glucose change: the difference between the pre-dialysis fasting plasma glucose (in mmol/L) measured at the end of the study period and the baseline value.
Number of Participants Who Permanently Discontinue the Study Intervention Due to an Adverse Event | 2 years
  This measure records participants who permanently stop receiving either the hemoperfusion or the continuous glucose infusion protocol specifically because of an adverse event, regardless of the event's severity or relationship assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- Blood Purification Center, Suzhou Hospital Affiliated to Anhui Medical University, Suzhou, Anhui, China

IPD SHARING:
Plan to Share IPD: Yes